CLINICAL TRIAL: NCT01922947
Title: Motivational Interviewing Integrated With Social Network Counseling for Teens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HM14479; 1R34DA032808-01A1 (NIH)
Record Dates: First submitted 2013-07-23; First posted 2013-08-14 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Substance Use
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Motivational Interviewing w/Social Network Counseling (Active Comparator): Motivational Interviewing integrated with Social Network Counseling, 20-minute session.
  Interventions: Behavioral: Active Control Condition
- Health Counseling (Sham Comparator)
  Interventions: Behavioral: Motivational Interviewing w/Social Network Counseling

INTERVENTIONS:
Behavioral: Motivational Interviewing w/Social Network Counseling — This is the active arm of the study.
  Arms: Health Counseling
Behavioral: Active Control Condition — 20-minute health counseling
  Arms: Motivational Interviewing w/Social Network Counseling

SUMMARY:
The purpose of this research is to test the feasibility and efficacy of a brief (one session) preventative intervention using motivational interviewing integrated with social network counseling for substance use among adolescent patients in a primary care setting. One hundred participants will be randomly assigned to either motivational interviewing integrated with social network counseling or attention control conditions. The motivational interviewing integrated with social network counseling condition is expected to show improvement when compared to the attention control condition.

ELIGIBILITY:
Inclusion Criteria:

* 14-18 years old
* Resident of Richmond VA or greater Richmond area
* Patient at Virginia Commonwealth University or Richmond City Department of Health

Exclusion Criteria:

* Ward of the state
* Not fluent in English
* Incapable of providing consent

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2012-08; Primary Completion 2014-11-30 (Actual); Study Completion 2014-11-30 (Actual)

PRIMARY OUTCOMES:
Effects of counseling on substance use factors in teens | Feb. 2015
  To assess the efficacy of motivational interviewing integrated with social network counseling compared to an attention control condition on substance use factors in teens assessed via self-report questionnaires at baseline, 1, 3, and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Mason, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States